CLINICAL TRIAL: NCT02851524
Title: Proof of Concept Study Concerning Vestibular Stimulation Using a New Method of Dynamic Posturography.
Acronym: POSTURODYN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: REVERCHON AOI 2015
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Vestibular Stimulation
MeSH Terms: interventions — Cytidine Diphosphate

ARMS (1):
- posturography (Experimental)
  Interventions: Other: posturography

INTERVENTIONS:
Other: posturography

SUMMARY:
Falls in the elderly population are a major public health problem because of their frequency and their consequences, notably in terms of dependence their cost to society. In most cases, balance disorders related to an impaired vestibular system are blamed, even though there is no formal evidence that this is the case.

Vestibular tests in routine otoneurological practice are based on the exploration of vestibulo-ocular or even vestibulo-cortical reflexes. They are not particularly suitable to screen for vestibular disorders in falls.

A prototype rocking chair has been developed to test psycho-vestibular pathways, defined as the pathways via which vestibular afferents are transported to the subject's conscience. Thanks to this apparatus, a stimulus of body movement will be generated, but with limited tactile, visual and proprioceptive afferents, in such a way that the vestibular system alone is able to indicate to subjects their position in space. The subject will be required to detect oscillatory movement, and then to distinguish between a vestibular stimulus and a pulsed auditory stimulus.

The study hypothesis is that the movement stimulation generated by our prototype will be sufficient to stimulate the vestibular system, which will manifest itself as a conscious sensation of movement and by a vestibulo-ocular reflex causing oculomotor manifestations.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* National health insurance cover
* Written consent
* Subjects able to understand simple instructions and packaging information and to provide informed consent

Exclusion Criteria:

* Vertigo, consciousness disorders, nausea or pain before the tests
* Bilateral deafness
* History of neurological, rheumatic or orthopaedic disease likely by itself to trigger a fall
* Psychiatric disorder likely to compromise participation.
* Personal history of falls of undetermined cause.
* Présence de saccades et/ou nystagmus en position statique
* Femme enceinte

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06-23 (Actual); Primary Completion 2017-04-21 (Actual); Study Completion 2017-04-21 (Actual)

PRIMARY OUTCOMES:
Cinematics of eye movements (amplitude and direction) evaluated by videonystagmography (VNG). | At Day 0

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Guyon M, Chea C, Laroche D, Fournel I, Baudet A, Toupet M, Bozorg Grayeli A. Measuring threshold and latency of motion perception on a swinging bed. PLoS One. 2021 Jul 9;16(7):e0252914. doi: 10.1371/journal.pone.0252914. eCollection 2021. PMID 34242212